CLINICAL TRIAL: NCT01489865
Title: A Phase I/II Study of ABT-888 in Combination With 5-fluorouracil and Oxaliplatin (Modified FOLFOX-6) in Patients With Metastatic Pancreatic Cancer
Brief Title: ABT-888 With Modified FOLFOX6 in Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 2009-608
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Pancreas cancer; Veliparib; oxaliplatin
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — veliparib; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (9):
- Phase 1: ABT-888 40mg (Cohort 1) (Experimental): ABT-888 orally at 40mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6 with 5-FU bolus mFOLFOX-6: Oxaliplatin 85 mg/M2 IV on Day 1 Leucovorin 400 mg/m2 IV on Day 1; 5-FU 400 mg/m2 IV bolus followed by 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
  Interventions: Drug: ABT-888; Drug: mFOLFOX-6
- Phase 1: ABT-888 60 mg (Cohort 2) (Experimental): ABT-888 orally at 60mg with mFOLFOX-6 twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
  Interventions: Drug: ABT-888; Drug: mFOLFOX-6
- Phase 1: ABT-888 80 mg (Cohort 3) (Experimental): ABT-888 orally at 80mg with mFOLFOX-6 twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
  Interventions: Drug: ABT-888; Drug: mFOLFOX-6
- Phase 1: ABT-888 100 mg (Cohort 4) (Experimental): ABT-888 orally at 100mg with mFOLFOX-6 twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
  Interventions: Drug: ABT-888; Drug: mFOLFOX-6
- Phase 1: ABT-888 150 mg (Cohort 5) (Experimental): ABT-888 orally at 150mg with mFOLFOX-6 twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
  Interventions: Drug: ABT-888; Drug: mFOLFOX-6
- Phase 1: ABT-888 200 mg (Cohort 6) (Experimental): ABT-888 orally at 200mg with mFOLFOX-6 twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
  Interventions: Drug: ABT-888; Drug: mFOLFOX-6
- Phase 1: ABT-888 250 mg (Cohort 7) (Experimental): ABT-888 orally at 250mg with mFOLFOX-6 twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
  Interventions: Drug: ABT-888; Drug: mFOLFOX-6
- Phase 1: ABT-888 300 mg (Cohort 8) (Experimental): ABT-888 orally at 300mg with mFOLFOX-6 twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
  Interventions: Drug: ABT-888; Drug: mFOLFOX-6
- Phase 2: ABT-888 at Recommended phase 2 dose (200mg) (Experimental): ABT-888 orally at 200mg with mFOLFOX-6 twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
  Interventions: Drug: ABT-888; Drug: mFOLFOX-6

INTERVENTIONS:
Drug: ABT-888 — ABT-888 in escalating doses twice a day for Days 1-7 of each 14-day cycle
  Other Names: veliparib
Drug: mFOLFOX-6 — Oxaliplatin 85 mg/M2 IV on Day 1 Leucovorin 400 mg/m2 IV on Day 1 5-FU 400 mg/m2 IV bolus followed by 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
  Other Names: 5-Fluorouracil; Eloxatin

SUMMARY:
People are being asked to participate in this study who have metastatic pancreatic cancer (cancer that has spread to other parts of the body).

The purpose of this study is to test the efficacy (effectiveness) of a new combination of drugs, ABT-888 and mFOLFOX-6 (modified 5-Fluorouracil and Oxaliplatin) for patients with metastatic pancreatic cancer.

ABT-888 inhibits an enzyme called "PARP" which helps to fix damaged DNA. By inhibiting this enzyme, ABT-888 prevents cancer cells from repairing the damage caused by the mFOLFOX-6, and will hopefully increase the killing of cancer cells, thus decreasing the tumors in your body.

DETAILED DESCRIPTION:
This is a single arm, open-label Phase I/II study to evaluate the clinical activity of the novel inhibitor of Poly(ADP-ribose) polymerase (PARP), ABT-888 with modified FOLFOX-6 (5-Fluorouracil plus oxaliplatin) in patients with metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven pancreatic adenocarcinoma with measurable disease
* A known BRCA-associate genetic mutation OR family history suggesting of a breast or ovarian cancer syndrome, as defined by one or more of the following:
* Personal or known family history of a deleterious (or indeterminate) mutation in the BRCA1, BRCA2, PALBB2, or one of the FANC genes.
* Personal history of breast cancer and one or more of the following:

  * Diagnosed ≤ 45 years old
  * Diagnosed at any age with ≥1 1st, 2nd, or 3rd degree relative with breast cancer ≤ 50 years old and/or ≥1st, 2nd, or 3rd relative with epithelial ovarian cancer at any age
  * Two primary breast cancer with the first diagnosed at ≤ 50 years old
  * Diagnosed ≤ 60 years old with triple negative breast cancer
  * Diagnosed at any age with ≥2 1st, 2nd, or 3rd degree relatives with breast cancer at any age
  * Diagnosed at any age with ≥2 1st, 2nd, or 3rd degree relatives with pancreatic cancer or aggressive prostate cancer (Gleason score ≥7) at any age
  * 1st, 2nd, or 3rd degree male relative with breast cancer
  * Ashkenazi Jewish descent
* Personal history of epithelial ovarian cancer
* Personal history of male breast cancer
* Personal history of pancreatic cancer and ≥2 1st, 2nd, or 3rd degree relatives with breast, epitherlial ovarian, pancreatic, or aggressive prostate cancer (Gleason score ≥7) at any age
* Age >= 18 years
* ECOG performance status 0-2
* Subjects with no brain metastases or a history of previously treated brain metastases who have been treated with surgery or stereotactic radiosurgery at least 4 weeks prior to enrollment and have a baseline MRI that shows no evidence of intercranial disease and have not had treatment with steroids within 1 week of study enrollment.
* Subjects may have received any number of prior therapies except prior therapy with a PARP inhibitor
* At least 14 days must have passed since all prior anti-cancer therapy
* At least 28 days must have passed since any prior antibody-based therapies
* At least 28 days must have passed since any prior investigational agent
* All patients must have completely recovered from all transient side effects related to prior therapies and any side effects that are expected to be more durable or permanent must have resolved to Grade 1
* Adequate hepatic, bone marrow and renal function
* Partial thromboplastin time must be </= 2 X upper limit of institution's normal range and INR < 2. Subjects on an anticoagulant must have a PTT </= 5 X upper limit of institution's normal range and INR < 5.
* Life expectancy > 12 weeks
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of treatment
* Subject must be capable of understanding and complying with parameters as outlined in protocol and able to sign and date the informed consent form
* Patients must have fully recovered from all effects of surgery.

Exclusion Criteria:

* Active severe infection, or known chronic infection with HIV, Hepatitis B virus or Hepatitis C virus
* Cardiovascular disease problems including unstable angina, therapy for life-threatening ventricular arrhythmia, or myocardial infarction, stroke, or congestive heart failure within the last 6 months
* Life-threatening visceral disease or other severe concurrent disease
* Women who are pregnant or breast-feeding
* Anticipated survival under 3 months
* The subject has had another active malignancy within the past 5 years except for cervical cancer in situ, in situ carcinoma of the bladder, or non-melanoma carcinoma of the skin.
* Active uncontrolled infection
* Symptomatic congestive heart failure
* Unstable angina pectoris or cardiac arrhythmia
* Psychiatric illness/ social situation that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-01-03 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2023-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pishvaian, MD PhD, Study Chair — Johns Hopkins University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: ABT-888 40mg (Cohort 1): ABT-888 orally at 40mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6 with 5-FU bolus:
  Oxaliplatin 85 mg/M2 IV on Day 1 Leucovorin 400 mg/m2 IVon Day 1; 5-FU 400 mg/m2 IV bolus followed by 2400 mg/m2 IV continuous infusion over 46 hoursDays 1-3
- Phase 1: ABT-888 60 mg (Cohort 2): ABT-888 orally at 60mg twice a day for Days 1-7 of each 14-day cycle. mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusionover 46 hours Days 1-3
- Phase 1: ABT-888 80 mg (Cohort 3): ABT-888 orally at 80 mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6:
  Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusionover 46 hours Days 1-3
- Phase 1: ABT-888 100 mg (Cohort 4): ABT-888 orally at 100mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6:
  Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusionover 46 hours Days 1-3
- Phase 1: ABT-888 150 mg (Cohort 5): ABT-888 orally at 150mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6:
  Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusionover 46 hours Days 1-3
- Phase 1: ABT-888 200 mg (Cohort 6); Phase 2: ABT-888 at Recommended Phase 2 Dose (200mg): ABT-888 orally at 200mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6:
  Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusionover 46 hours Days 1-3
- Phase 1: ABT-888 250 mg (Cohort 7): ABT-888 orally at 250mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6:
  Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusionover 46 hours Days 1-3
- Phase 1: ABT-888 300 mg (Cohort 8): ABT-888 orally at 300mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6:
  Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusionover 46 hours Days 1-3
Period: Overall Study
Arm/Group | Phase 1: ABT-888 40mg (Cohort 1) | Phase 1: ABT-888 60 mg (Cohort 2) | Phase 1: ABT-888 80 mg (Cohort 3) | Phase 1: ABT-888 100 mg (Cohort 4) | Phase 1: ABT-888 150 mg (Cohort 5) | Phase 1: ABT-888 200 mg (Cohort 6) | Phase 1: ABT-888 250 mg (Cohort 7) | Phase 1: ABT-888 300 mg (Cohort 8) | Phase 2: ABT-888 at Recommended Phase 2 Dose (200mg)
Started | 6 | 3 | 3 | 3 | 3 | 7 | 6 | 0 | 33
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 6 | 3 | 3 | 3 | 3 | 7 | 6 | 0 | 32
Not completed — Progression of Disease | 4 | 2 | 2 | 3 | 1 | 6 | 3 | 0 | 23
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 5
Not completed — Death | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Not completed — Shifted | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: ABT-888 60 mg (Cohort 2): ABT-888 orally at 60mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/M2 IV on Day 1 Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 1: ABT-888 80 mg (Cohort 3): ABT-888 orally at 80mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/M2 IV on Day 1 Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 1: ABT-888 100 mg (Cohort 4): ABT-888 orally at 100mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/M2 IV on Day 1 Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 1: ABT-888 150 mg (Cohort 5): ABT-888 orally at 150mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/M2 IV on Day 1 Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 1: ABT-888 200 mg (Cohort 6); Phase 2: ABT-888 atRecommended Phase 2 Dose (200mg): ABT-888 orally at 200mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/M2 IV on Day 1 Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 1: ABT-888 250 mg (Cohort 7): ABT-888 orally at 250mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/M2 IV on Day 1 Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Total: Total of all reporting groups
Arm/Group | Phase 1: ABT-888 40mg (Cohort 1) | Phase 1: ABT-888 60 mg (Cohort 2) | Phase 1: ABT-888 80 mg (Cohort 3) | Phase 1: ABT-888 100 mg (Cohort 4) | Phase 1: ABT-888 150 mg (Cohort 5) | Phase 1: ABT-888 200 mg (Cohort 6) | Phase 1: ABT-888 250 mg (Cohort 7) | Phase 2: ABT-888 atRecommended Phase 2 Dose (200mg) | Total
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 7 | 6 | 33 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 3 | 2 | 0 | 5 | 4 | 20 | 39
  >=65 years | 3 | 1 | 0 | 1 | 3 | 2 | 2 | 13 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 17 | 27
  Male | 4 | 2 | 2 | 1 | 2 | 5 | 5 | 16 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 6 | 3 | 3 | 2 | 3 | 7 | 6 | 30 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 7 | 11
  White | 6 | 2 | 3 | 2 | 3 | 5 | 5 | 23 | 49
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Dose Limiting Toxicities
Description: Protocol defined events that are definitely, possibly or probably related to one or both agents and have occurred in the first cycle of therapy. Applies only to patients in the Phase I portion of the study.
Time Frame: 28 days
Measure: Number; unit: Dose Limiting Toxicities
Groups:
- Phase 1: ABT-888 40mg (Cohort 1): ABT-888 orally at 40mg twice a day for Days 1-7 of each 14-day cycle with 5-FU bolus mFOLFOX-6: Oxaliplatin 85 mg/M2 IVon Day 1 Leucovorin 400 mg/m2 IVon Day 1; 5-FU 400 mg/m2 IV bolus followed by 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 1: ABT-888 100 mg (Cohort 4): ABT-888 orally at 100mg twice a day for Days 1-7of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/M2 IV on Day 1 Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 1: ABT-888 150 mg (Cohort 5): ABT-888 orally at 150mg twice a day for Days 1-7of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusionover 46 hours Days 1-3
- Phase 1: ABT-888 200 mg (Cohort 6): ABT-888 orally at 200mg with mFOLFOX-6 twice a day for Days 1-7of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 2400 mg/m2 IV continuous infusionover 46 hours Days 1-3
Arm/Group | Phase 1: ABT-888 40mg (Cohort 1) | Phase 1: ABT-888 60 mg (Cohort 2) | Phase 1: ABT-888 80 mg (Cohort 3) | Phase 1: ABT-888 100 mg (Cohort 4) | Phase 1: ABT-888 150 mg (Cohort 5) | Phase 1: ABT-888 200 mg (Cohort 6) | Phase 1: ABT-888 250 mg (Cohort 7)
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 7 | 6
Dose Limiting Toxicities | 3 | 0 | 0 | 0 | 0 | 0 | 4

2. Primary Outcome: Phase II: Objective Response Rate (ORR)
Description: Number of Participants in Phase II with a Complete response and Partial response as determined by RECIST 1.1.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- ABT-888 and mFOLFOX-6 Phase II: ABT-888 orally at escalating does in Phase I and then at recommended phase II dose with standard mFOLFOX-6
  ABT-888 and mFOLFOX-6: ABT-888 in escalating doses twice a day for Days 1-7 of each 14-day cycle Oxaliplatin 85 mg/M2 IV on Day 1 Leucovorin 400 mg/m2 IV on Day 1 5-FU 400 mg/m2 IV bolus followed by 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
Arm/Group | ABT-888 and mFOLFOX-6 Phase II
Number analyzed (Participants) | 33
Participants | 4

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the number of patients with a complete response, partial response, or stable disease at 6 months per Recist 1.1.
Time Frame: 6 months
Population: response-evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: ABT-888 60 mg (Cohort 2): ABT-888 orally at 60mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; ; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 1: ABT-888 80 mg (Cohort 3): ABT-888 orally at 80mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 1: ABT-888 100 mg (Cohort 4): ABT-888 orally at 100mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 1: ABT-888 150 mg (Cohort 5): ABT-888 orally at 150mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 1: ABT-888 200 mg (Cohort 6): ABT-888 orally at 200mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 1: ABT-888 250 mg (Cohort 7): ABT-888 orally at 250mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 2: ABT-888 at Recommended Phase 2 Dose (200mg): ABT-888 orally at 200mg with mFOLFOX-6 twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6:
  Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
Arm/Group | Phase 1: ABT-888 40mg (Cohort 1) | Phase 1: ABT-888 60 mg (Cohort 2) | Phase 1: ABT-888 80 mg (Cohort 3) | Phase 1: ABT-888 100 mg (Cohort 4) | Phase 1: ABT-888 150 mg (Cohort 5) | Phase 1: ABT-888 200 mg (Cohort 6) | Phase 1: ABT-888 250 mg (Cohort 7) | Phase 2: ABT-888 at Recommended Phase 2 Dose (200mg)
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 7 | 6 | 33
Participants | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 5

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the number of days from enrollment to progression or death, whichever occurred first.
Time Frame: up to 114 months
Measure: Median (Full Range); unit: days
Groups:
- Phase 1: ABT-888 60 mg (Cohort 2): ABT-888 orally at 60mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
- Phase 2: ABT-888 at Recommended Phase 2 Dose (200mg): ABT-888 orally at 200mg twice a day for Days 1-7 of each 14-day cycle with mFOLFOX-6: Oxaliplatin 85 mg/m2 IV on Day 1; Leucovorin 400 mg/m2 IV on Day 1; 5-FU 2400 mg/m2 IV continuous infusion over 46 hours Days 1-3
Arm/Group | Phase 1: ABT-888 40mg (Cohort 1) | Phase 1: ABT-888 60 mg (Cohort 2) | Phase 1: ABT-888 80 mg (Cohort 3) | Phase 1: ABT-888 100 mg (Cohort 4) | Phase 1: ABT-888 150 mg (Cohort 5) | Phase 1: ABT-888 200 mg (Cohort 6) | Phase 1: ABT-888 250 mg (Cohort 7) | Phase 2: ABT-888 at Recommended Phase 2 Dose (200mg)
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 7 | 6 | 33
days | 126.5 [65 to 509] | 49 [42 to 58] | 159 [91 to 948] | 77 [56 to 106] | 132 [37 to 671] | 148 [33 to 209] | 60.5 [49 to 122] | 102 [15 to 3431]

5. Secondary Outcome: Overall Survival
Description: The number of days from enrollment until death or last contact. Patients who were alive at the time of analysis were censored at their last contact.
Time Frame: up to 114 months
Measure: Median (Full Range); unit: days
Arm/Group | Phase 1: ABT-888 40mg (Cohort 1) | Phase 1: ABT-888 60 mg (Cohort 2) | Phase 1: ABT-888 80 mg (Cohort 3) | Phase 1: ABT-888 100 mg (Cohort 4) | Phase 1: ABT-888 150 mg (Cohort 5) | Phase 1: ABT-888 200 mg (Cohort 6) | Phase 1: ABT-888 250 mg (Cohort 7) | Phase 2: ABT-888 at Recommended Phase 2 Dose (200mg)
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 7 | 6 | 33
days | 153 [89 to 750] | 89 [58 to 169] | 325 [159 to 948] | 294 [146 to 320] | 211 [37 to 671] | 176 [104 to 319] | 145.5 [49 to 336] | 260 [15 to 3431]

ADVERSE EVENTS:
Time Frame: From the time of study drug administration until 30 days following discontinuation of study drug administration, up to 10 years.
Arm/Group | Phase 1: ABT-888 40mg (Cohort 1) | Phase 1: ABT-888 60 mg (Cohort 2) | Phase 1: ABT-888 80 mg (Cohort 3) | Phase 1: ABT-888 100 mg (Cohort 4) | Phase 1: ABT-888 150 mg (Cohort 5) | Phase 1: ABT-888 200 mg (Cohort 6) | Phase 1: ABT-888 250 mg (Cohort 7) | Phase 2: ABT-888 at Recommended Phase 2 Dose (200mg)
All-Cause Mortality (participants affected / at risk) | 6/6 | 3/3 | 3/3 | 3/3 | 3/3 | 7/7 | 6/6 | 30/33
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/3 | 0/3 | 0/3 | 2/3 | 0/7 | 3/6 | 12/33
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 3/3 | 3/3 | 3/3 | 6/6 | 4/7 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: ABT-888 40mg (Cohort 1) (N=6) | Phase 1: ABT-888 60 mg (Cohort 2) (N=3) | Phase 1: ABT-888 80 mg (Cohort 3) (N=3) | Phase 1: ABT-888 100 mg (Cohort 4) (N=3) | Phase 1: ABT-888 150 mg (Cohort 5) (N=3) | Phase 1: ABT-888 200 mg (Cohort 6) (N=7) | Phase 1: ABT-888 250 mg (Cohort 7) (N=6) | Phase 2: ABT-888 at Recommended Phase 2 Dose (200mg) (N=33)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — complete heart block
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Pneumonia
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Gram Negative bacteremia
Sepsis (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Liver enzymes elevated
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: ABT-888 40mg (Cohort 1) (N=6) | Phase 1: ABT-888 60 mg (Cohort 2) (N=3) | Phase 1: ABT-888 80 mg (Cohort 3) (N=3) | Phase 1: ABT-888 100 mg (Cohort 4) (N=3) | Phase 1: ABT-888 150 mg (Cohort 5) (N=3) | Phase 1: ABT-888 200 mg (Cohort 6) (N=6) | Phase 1: ABT-888 250 mg (Cohort 7) (N=7) | Phase 2: ABT-888 at Recommended Phase 2 Dose (200mg) (N=33)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 1 (1) | 3 (4)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 4 (6) | 2 (2) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 2 (3) | 2 (2) | 9 (10)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 3 (3) | 3 (4) | 2 (2) | 4 (4) | 4 (6) | 25 (38)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (5) | 0 (0) | 3 (4) | 2 (2) | 14 (18)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 4 (5) | 3 (3) | 2 (4) | 3 (4) | 2 (3) | 4 (5) | 3 (4) | 23 (29)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 3 (3)
Pain (General disorders) | 2 (3) | 1 (2) | 1 (1) | 1 (2) | 2 (3) | 4 (5) | 1 (1) | 2 (3)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (10)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (10)
Lymphocyte count decreased (Investigations) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (7) | 0 (0) | 1 (1) | 1 (2) | 1 (4) | 3 (9) | 3 (5) | 7 (16)
Platelet count decreased (Investigations) | 3 (3) | 0 (0) | 1 (11) | 0 (0) | 2 (6) | 3 (4) | 3 (7) | 2 (5)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
White blood cell decreased (Investigations) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 3 (5) | 2 (7)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 12 (14)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Dysesthesia (Nervous system disorders) | 2 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 6 (6)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Paresthesia (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 9 (10)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Hypertension (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT01489865/Prot_SAP_000.pdf